CLINICAL TRIAL: NCT02813382
Title: Intrathecal 60mg Prilocaine, Hyperbaric 40mg 9-chloroprocaine and 10.5mg Bupivacaine Each With Added Sufentanil (2µg) for Elective Ambulatory Umbilical and Unilateral Inguinal Herniorrhaphy
Brief Title: Spinal Anesthesia for Outpatient Abdominal Wall Surgery: Comparison of Bupivacaine, 2-chloroprocaine and Prilocaine
Acronym: spinal
Status: Completed | Type: Observational
Sponsor: AZ St.-Dimpna Geel (Other)
Responsible Party: Principal Investigator, Ben Gys, md, AZ St.-Dimpna Geel
Other Study IDs: Spinal-001
Record Dates: First submitted 2016-06-19; First posted 2016-06-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia, Spinal; Ambulatory Surgical Procedures; Hernia, Inguinal; Hernia, Umbilical
Keywords: bupivacaine; prilocaine; 2-chloroprocaine
MeSH Terms: conditions — Hernia, Inguinal; Hernia, Umbilical | interventions — Bupivacaine; Prilocaine; chloroprocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- B-group: Spinal anesthesia was performed using 10.5mg bupivacaine with added sufentanil (2µg).
  Interventions: Drug: Bupivacaine
- C-group: Spinal anesthesia was performed using 40mg hyperbaric 2-chloroprocaïne with added sufentanil (2µg).
  Interventions: Drug: Chloroprocaine
- P-group: Spinal anesthesia was performed using 60mg prilocaïne with added sufentanil (2µg).
  Interventions: Drug: Prilocaine

INTERVENTIONS:
Drug: Bupivacaine — Spinal anesthesia was performed using 10.5mg bupivacaine with added sufentanil (2µg).
  Groups: B-group
Drug: Prilocaine — Spinal anesthesia was performed using 60mg prilocaïne with added sufentanil (2µg).
  Groups: P-group
Drug: Chloroprocaine — Spinal anesthesia was performed using 40mg hyperbaric 2-chloroprocaïne with added sufentanil (2µg).
  Other Names: 2-chloroprocaine
  Groups: C-group

SUMMARY:
Considering fast-track principles, an ideal spinal anesthetic should have minimal complications and above all fast recovery so reducing in-hospital stay.

Between 1/8/2015 and 1/1/2016, a total of 101 patients attending the surgeon's practice with an umbilical or unilateral inguinal hernia and no contra-indications for surgery were included in this study. Patients were given 10.5mg bupivacaine (B-group), 40mg hyperbaric 2-chloroprocaïne (C-group) or 60mg prilocaïne (P-group), each with added sufentanil (2µg). Motor block was assessed using the Bromage scale. Sensory block was measured by determining the peak level dermatome. Intraoperative hemodynamic parameters were listed. Resolution of sensory and motor block, time to void and home readiness were defined as clinical endpoints.

DETAILED DESCRIPTION:
Open inguinal and umbilical hernia repair are two of the most performed interventions in day-care surgery. Fast-track surgery implies a swift and effective form of anesthesia which is easy to carry out, has few side-effects and is quickly reversed.

Spinal anesthesia has proven to be a safe method to ensure adequate analgesia for patients undergoing elective open abdominal wall surgery as the need and side-effects of general anesthesia are avoided. During many years, a variety of intrathecal products alongside a plethora of adjuvants have been evaluated.

Three different types of spinal anesthetic products already used in routine care were compared: hyperbaric 9-chloroprocaïne (Ampres®, Nordic Pharma), bupivacaine (Marcaine®, AstraZeneca) and prilocaine (Tachipri®, Nordic Pharma).

Between 1/8/2015 and 1/1/2016, a total of 101 patients attending the surgeon's practice with an umbilical or unilateral inguinal hernia and no contra-indications for surgery were included in this study. Local ethical committee approval (EC0G099 - AZ Sint Dimpna, Geel, Belgium) and individual written informed consent was obtained. Surgical procedures were performed by 2 surgeons (TL and TG). The hernia was diagnosed clinically and/or by ultrasonography. Patients were preoperatively informed about the details concerning surgery and anesthesiology.

All patients were hospitalized on the day of surgery following standard preoperative instructions. Spinal anesthesia was performed by 6 different anesthesiologists. Patients with contraindications for spinal anesthesia were excluded: INR (international normalized ratio) > 1.2, thrombocytopenia (<75.000/µl), symptomatic neurological disease and proven allergy for local anesthetic. All patients received 1g of cefazolin (following standard guidelines for antibiotic prophylaxis of surgical wounds).

Patient's baseline features were listed: gender, age, Body Mass Index (BMI), Anesthesiologists Physical Status classification (ASA classification), their position at the moment of intrathecal infusion (sitting up or lateral decubitus) and type and length of surgery. Open inguinal herniorrhaphy was performed following the Liechtenstein technique as described by Chastan. For the treatment of an umbilical hernia, a polypropylene-ePTFE hernia patch (Ventralex™, BARD®) was used .

Patients were given 10.5mg bupivacaine (B-group), 40.0mg of hyperbaric 2-chloroprocaïne (C-group) or 60.0mg prilocaïne (P-group), each in combination with sufentanil (2.0µg).

All patients with pre-existing hypotension (<120/80) were administered 5.0mg of ephedrine and 0.2mg of glycopyrroniumbromide IV upon entering the operation theater through a standard peripheral catheter. Regular monitoring was used during the procedure: electronic blood pressure monitoring, pulse oximetry and 3-lead electrocardiogram. Hemodynamic anomalies were listed: hypotension (systolic pressure <75% of baseline value), bradycardia (pulse <60/min) and desaturation (<92% without oxygen).

Under sterile conditions, local anesthesia of the skin of the lower back was performed (using 1% 3cc lidocaine). Afterwards, puncture of the arachnoid mater (using a 25G Sprottle Needle) was performed at the L2-L3 interspace and the predetermined product instilled. This procedure was performed sitting-up or in dorsolateral decubitus (in inguinal hernia repair lying on the ipsilateral side when using prilocaine or bupivacaine and on the contralateral side when using hyperbaric 2-chloroprocaine). Patients who received their spinal block in the sitting up position were instantly put in the dorsolateral position after the injection (side again depending on the product and type of surgery as described above). Regardless of these proceedings, all patients receiving 9-chloroprocaine were put in the reverse Trendelenburg position (approximately 20°) for 2 minutes immediately after infusion.

After injection, sensory and motor block assessment was performed and listed on predetermined moments: 1, 3, 30 minutes after infusion and from then on every 15 minutes until spontaneous voiding (>200ml) was achieved. Sensory block was evaluated from toe to head at the surgical side using the loss of sensation to cold fluids (ether). Motor block was assessed using the Bromage scale.

During surgery, hypotension (systolic pressure <75% of baseline value) was treated with ephedrine and bradycardia with atropine or ephedrine. Patients who suffered from desaturation (blood oxygen saturation <92%) received oxygen through a standard face mask starting at 2l/min. Fentanyl 25 to 100µg was given when pain was felt by the patient. If insufficient analgesia was achieved (insufficient sensory block), general anesthesia was initiated. Intraoperative IV analgesia consisted of standard postoperative pain medication (taradyl and perfusalgan). If there was a history of duodenal ulcus, kidney insufficiency and/or intolerance for NSAIDs, taradyl was replaced with dynastat.

Postoperatively, all patients were transferred to the Post-Anesthesia Care Unit (PACU), where they received standard postoperative analgesia (paracetamol 1g IV and/or taradyl 30mg IV). If insufficient, fentanyl was administered. Postoperative nausea and vomiting (PONV) was treated with alizapride and ondansetron. After a minimum stay of 90 minutes, signs of regression of the motor block (Bromage scale) and normal hemodynamic parameters, patients were transferred to the day-care hospital for further recovery.

Resolution of sensory and motor blockage, time to void and home readiness (spontaneous voiding, ability to walk without assistance, the absence of nausea or vomiting and stable hemodynamic parameters) were defined as clinical endpoints. Pain experienced at the day-care hospital was managed with oral paracetamol (500mg) and/or ibuprofen (600mg), after determination of a Visual Analog Scale for Pain (VAS).

All data was analyzed using IBM SPSS statistical software version 23 and Microsoft Excel 2010. Comparison of continuous variables was performed using the F-test and posthoc analysis . Categorical variables were compared by means of a chi-square test. A P-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* unilateral open inguinal or umbilical hernia repair
* capable to understand the risks and commitment associated with the surgery and anesthesia

Exclusion Criteria:

* concomittant surgical of non-surgical procedure
* no agreement to informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 105 consecutive patients undergoing elective unilateral open inguinal or umbilical hernia repair.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time to void | up to 24hours after surgery
  Postoperative spontaneous voiding (>200ml).

SECONDARY OUTCOMES:
in hospital time | up to 24hours after surgery
time from spinal anesthesia to ready-to-cut | an average of 3 minutes
time from spinal anesthesia to start of surgery | an average of 3 minutes
time to T6 | 1 hour
  Time to reach sensory block at the T6 dermatome after intrathecal infusion.
time to T10 | 1 hour
  Time to reach sensory block at the T10 dermatome after intrathecal infusion.
time to onset of peak sensory level block | an average of 60 minutes
peak sensory level (dermatome) | an average of 60 minutes
  Peak sensory block height (according to dermatomes).

CONTACTS AND LOCATIONS:
Overall Officials: Ben Gys, md, Principal Investigator — AZ Sint Dimpna, Geel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Goldblum E, Atchabahian A. The use of 2-chloroprocaine for spinal anaesthesia. Acta Anaesthesiol Scand. 2013 May;57(5):545-52. doi: 10.1111/aas.12071. Epub 2013 Jan 16. PMID 23320599
- [Result] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878
- [Result] Forster JG. Short-acting spinal anesthesia in the ambulatory setting. Curr Opin Anaesthesiol. 2014 Dec;27(6):597-604. doi: 10.1097/ACO.0000000000000126. PMID 25211156
- [Result] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Result] Akcaboy ZN, Akcaboy EY, Mutlu NM, Serger N, Aksu C, Gogus N. Spinal anesthesia with low-dose bupivacaine-fentanyl combination: a good alternative for day case transurethral resection of prostrate surgery in geriatric patients. Rev Bras Anestesiol. 2012 Nov-Dec;62(6):753-61. doi: 10.1016/S0034-7094(12)70176-9. PMID 23176984